CLINICAL TRIAL: NCT03704298
Title: A Phase 1/2 Multi-center Study Evaluating the Safety and Efficacy of Axicabtagene Ciloleucel in Combination With Utomilumab in Subjects With Relapsed/Refractory Large B-Cell Lymphoma
Brief Title: Safety and Efficacy of Axicabtagene Ciloleucel in Combination With Utomilumab in Adults With Refractory Large B-cell Lymphoma
Acronym: ZUMA-11
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Development program terminated
Sponsor: Kite, A Gilead Company (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KTE-C19-111
Record Dates: First submitted 2018-10-10; First posted 2018-10-12 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Relapsed/Refractory Large B-cell Lymphoma
MeSH Terms: conditions — Recurrence | interventions — Cyclophosphamide; fludarabine; axicabtagene ciloleucel; utomilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1: Cohort 1: Axicabtagene Ciloleucel + Utomilumab 10 mg (Experimental): Participants will receive cyclophosphamide 500 mg/m^2/day intravenously (IV) and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-cluster of differentiation (CD) 19 chimeric antigen receptor (CAR) transduced autologous T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells will be administered. Participants also will receive utomilumab 10 mg on Day 1, IV infusion, once every 4 weeks (Q4W) for 6 months or until progressive disease, whichever came first.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Axicabtagene Ciloleucel; Biological: Utomilumab
- Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg (Experimental): Participants will receive cyclophosphamide 500 mg/m^2/day IV and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR transduced autologous T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells will be administered. Participants also will receive utomilumab 30 mg on Day 1, IV infusion, Q4W for 6 months or until progressive disease, whichever came first.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Axicabtagene Ciloleucel; Biological: Utomilumab
- Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg (Experimental): Participants will receive cyclophosphamide 500 mg/m^2/day IV and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR transduced autologous T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells will be administered. Participants also will receive utomilumab 100 mg on Day 1, IV infusion, Q4W for 6 months or until progressive disease, whichever came first.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Axicabtagene Ciloleucel; Biological: Utomilumab
- Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg (Experimental): Participants will receive cyclophosphamide 500 mg/m^2/day IV and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR transduced autologous T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells will be administered. Participants also will receive utomilumab 200 mg on Day 1, IV infusion, Q4W for 6 months or until progressive disease, whichever came first.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Axicabtagene Ciloleucel; Biological: Utomilumab
- Phase 1: Cohort 5: Axicabtagene Ciloleucel + Utomilumab 400 mg (Experimental): Participants will receive cyclophosphamide 500 mg/m^2/day IV and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR transduced autologous T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells will be administered. Participants also will receive utomilumab 400 mg on Day 1, IV infusion, Q4W for 6 months or until progressive disease, whichever came first.
  However, as the study was early terminated, no participants were enrolled in Cohort 5 of the study.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Axicabtagene Ciloleucel; Biological: Utomilumab
- Phase 2: Axicabtagene Ciloleucel + Utomilumab (Experimental): Participants will receive cyclophosphamide 500 mg/m^2/day IV and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel and utomilumab based on the dose and schedule selected to move forward from the Phase 1 portion of the study as recommended by the internal safety review team.
  However, as the study was early terminated, no participants were enrolled in Phase 2 of the study.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Axicabtagene Ciloleucel; Biological: Utomilumab

INTERVENTIONS:
Drug: Cyclophosphamide — Administered according to package insert
Drug: Fludarabine — Administered according to package insert
Biological: Axicabtagene Ciloleucel — A single infusion of chimeric antigen receptor (CAR)-transduced autologous T cells administered intravenously
  Other Names: Yescarta®
Biological: Utomilumab — Administered as an IV infusion

SUMMARY:
The primary objectives of this study are:

Phase 1: To evaluate the safety of axicabtagene ciloleucel in combination with utomilumab and to identify the most appropriate dose and timing of utomilumab to carry forward into Phase 2

Phase 2: To evaluate the efficacy of axicabtagene ciloleucel and utomilumab as measured by complete response rate in participants with refractory large B-cell lymphoma

DETAILED DESCRIPTION:
This study was intended to be a Phase 1/2. Enrollment was stopped prior to completion of Phase 1 portion of the study based on the sponsor's decision to end the program. No participants were enrolled in Phase 1 Cohort 5 and Phase 2.

After the study ends, participants who received an infusion of axicabtagene ciloleucel and utomilumab will complete the remainder of the 15-year follow-up assessments in a separate Long-term Follow-up study, KT-US-982-5968 (NCT05041309).

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically proven large B-cell lymphoma including the following types:

  * Diffuse large B cell lymphoma (DLBCL) not otherwise specified Activated B cell / Germinal center B cell (ABC/GCB).
  * High grade B-cell lymphoma (HGBCL) with or without MYC and BCL2 and/or BCL6 rearrangement.
  * DLBCL arising from follicular lymphoma.
  * T cell/histiocyte rich large B-cell lymphoma.
  * DLBCL associated with chronic inflammation.
  * Primary cutaneous DLBCL, leg type.
  * Epstein-Barr virus (EBV) + DLBCL
* Relapsed or chemotherapy-refractory disease, defined as one or more of the following:

  * No response to first-line therapy (primary refractory disease); individuals who are intolerant to first-line systemic chemotherapy are excluded

    * Progressive disease (PD) as best response to first-line therapy.
    * Stable disease (SD) as best response after at least 4 cycles of first-line therapy (eg, 4 cycles of R-CHOP) with SD duration no longer than 6 months from last dose of therapy.
  * No response to second or greater lines of therapy.

    * PD as best response to most recent therapy regimen.
    * SD as best response after at least 2 cycles of last line of therapy with SD duration no longer than 6 months from last dose of therapy OR
  * Refractory post-autologous stem cell transplant (ASCT).

    * Disease progression or relapsed 12 months after ASCT (must have biopsy proven recurrence in relapsed individual).
    * if salvage therapy is given post-ASCT, the individual must have had no response to or relapsed after the last line of therapy .
  * Relapsed or refractory LBCL including DLBCL, Transformed follicular lymphoma (TFL), and HGBCL after 2 or more lines of systemic therapy that is defined by and aligns with currently approved indication:

    * Relapsed disease after 2 or more lines of systemic therapy.
    * Best response that is less than a complete response to second or greater line of systemic therapy.
* At least 1 measurable lesion according to the Lugano Classification. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy.
* Individual must have received adequate prior therapy including at a minimum:

  * Anti-cluster of differentiation (CD) 20 monoclonal antibody unless investigator determines that tumor is CD20-negative, and
  * An anthracycline containing chemotherapy regimen.
* No radiographic evidence, suspicion and/or history of central nervous system (CNS) involvement of lymphoma.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Absolute neutrophil count (ANC) ≥ 1000/μL.
* Platelet count ≥ 75,000/μL.
* Absolute lymphocyte count ≥ 100/μL.
* Adequate renal, hepatic, pulmonary, and cardiac function defined as:

  * Creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 mL/min.
  * Serum alanine aminotransferase/aspartate aminotransferase (ALT/AST) ≤ 2.5 upper limit of normal (ULN).
  * Total bilirubin ≤ 1.5 mg/dL, except in individuals with Gilbert's syndrome.
  * Cardiac ejection fraction ≥ 50% and no evidence of pericardial effusion within 180 days provided the individual did not receive an anthracycline-based treatment or experience a cardiac event or change in performance status.
  * No clinically significant pleural effusion.
  * Baseline oxygen saturation > 92% on room air.

Key Exclusion Criteria:

* Histologically proven primary mediastinal B-cell lymphoma (PMBCL).
* History of Richter's transformation of chronic lymphocytic lymphoma (CLL).
* Prior chimeric antigen receptor therapy or other genetically modified T-cell therapy.
* History of severe, immediate hypersensitivity reaction attributed to aminoglycosides.
* History of human immunodeficiency virus (HIV) infection or acute or chronic active hepatitis B or C infection. Individuals with history of hepatitis infection must have cleared their infection as determined by standard serological and genetic testing per current Infectious Diseases Society of America (IDSA) guidelines or applicable country guidelines.
* Individuals with detectable cerebrospinal fluid malignant cells, brain metastases, or a history of CNS lymphoma.
* History or presence of CNS disorder, such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
* Individuals with cardiac atrial or cardiac ventricular lymphoma involvement.
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment.
* Requirement for urgent therapy due to tumor mass effects (eg, blood vessel compression, bowel obstruction, or transmural gastric involvement.
* Primary immunodeficiency.
* History of autoimmune disease (eg, Crohn's, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years. Individuals with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone and individuals with controlled type 1 diabetes mellitus on a stable insulin regimen may be eligible for this study.
* History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months of enrollment
* Any medical condition likely to interfere with assessment of safety or efficacy of study treatment
* Autologous stem cell transplant within 6 weeks of planned enrollment
* Prior organ transplantation including prior allogeneic stem cell transplant (SCT)
* Use of any standard or experimental anti-cancer therapy within 2 weeks prior to enrollment, including cytoreductive therapy and radiotherapy, immunotherapy, or cytokine therapy (except for erythropoietin) Prior treatment with PD-L1 inhibitor, PD-1 inhibitor, anti-CTLA4, anti-CD137 (4-1BB), anti-OX40 or other immune checkpoint blockade or activator therapy
* History of idiopathic pulmonary fibrosis, organizing pneumonia (eg, bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis per chest computed tomography (CT) scan at screening. History of radiation pneumonitis in the radiation field (fibrosis) is allowed.
* In the investigator's judgment, the individual is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (5):
- United States (5):
  - Stanford Cancer Institute, Palo Alto, California
  - UCLA Hematology/ Oncology, Santa Monica, California
  - Moffitt Cancer Center, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy/
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy/

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KTE-C19-111

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. This study was planned to be conducted in 2 parts: Phase 1 and Phase 2. Phase 1 was to be of 5 cohorts. Due to early termination of the study, Cohort 5 and Phase 2 were not conducted and no participants were enrolled in these cohorts. Results are reported only for Phase 1: Cohorts 1-4 of the study.
Pre-assignment Details: 17 participants were screened.
Groups:
- Phase 1: Cohort 1: Axicabtagene Ciloleucel + Utomilumab 10 mg: Participants received cyclophosphamide 500 mg/m^2/day intravenously (IV) and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-cluster of differentiation (CD)19 chimeric antigen receptor (CAR) transduced autologous T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells was administered. Participants also received utomilumab 10 mg on Day 1, IV infusion, once every 4 weeks (Q4W) for 6 months or until progressive disease, whichever came first.
- Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg: Participants received cyclophosphamide 500 mg/m^2/day IV and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR transduced autologous T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells was administered. Participants also received utomilumab 30 mg on Day 1, IV infusion, Q4W for 6 months or until progressive Disease, whichever came first.
- Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg: Participants received cyclophosphamide 500 mg/m^2/day IV and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR transduced autologous T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells was administered. Participants also received utomilumab 100 mg on Day 1, IV infusion, Q4W for 6 months or until progressive Disease, whichever came first.
- Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg: Participants received cyclophosphamide 500 mg/m^2/day IV and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR transduced autologous T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells was administered. Participants also received utomilumab 200 mg on Day 1, IV infusion, Q4W for 6 months or until progressive Disease, whichever came first.
Period: Overall Study
Arm/Group | Phase 1: Cohort 1: Axicabtagene Ciloleucel + Utomilumab 10 mg | Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg | Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg | Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg
Started | 5 | 4 | 3 | 3
Completed | 0 | 0 | 0 | 0
Not Completed | 5 | 4 | 3 | 3
Not completed — Death | 3 | 1 | 1 | 0
Not completed — Rollover to Long-term Follow-up Study Criteria | 1 | 2 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Developed Other Infection Before Starting the Treatment | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set is defined as all participants treated with any dose of axicabtagene ciloleucel.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Cohort 1: Axicabtagene Ciloleucel + Utomilumab 10 mg | Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg | Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg | Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 1 | 1 | 7
  >=65 years | 0 | 1 | 2 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (8.0) | 66 (9.6) | 64.0 (8.7) | 69.0 (10.6) | 63 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 0 | 5
  Male | 2 | 1 | 1 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 3 | 2 | 3 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 1 | 3 | 2 | 2 | 8
  More than one race | 1 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Percentage of Participants Experiencing Adverse Events Defined as Dose Limiting Toxicities (DLTs)
Description: DLTs are study drug-related events with onset within first 28 days following infusion of axicabtagene ciloleucel or utomilumab:
  * Grade (GR) 4 hematologic toxicity lasting more than 30 days (except lymphopenia or B-cell aplasia)
  * All study drug-related GR 3 lasting for > 7 days or 4 non-hematologic toxicities regardless of duration (except: aphasia/dysphasia or confusion/cognitive disturbance which resolves to at least GR 1 within 2 weeks or baseline within 4 weeks, fever of any grade, immediate study drug-related hypersensitivity reactions within 2 hours of drug infusion that are reversible to grade 2 or less within 24 hours, renal toxicity which requires dialysis for ≤ 7 days, intubation for airway protection if ≤ 7 days, tumor lysis syndrome, grade 3 liver function test elevation, provided there is resolution to ≤ GR 2 within 14 days, grade 4 transient serum hepatic enzyme abnormalities provided there is resolution to ≤ GR 3 within < 72 hours, grade 3 nausea and/or anorexia).
Time Frame: Up to 28 days
Population: The DLT evaluable set was defined as participants in each Phase 1 cohort who received the target axicabtagene ciloleucel dose and were followed for at least 28 days after the first utomilumab infusion or who received axicabtagene ciloleucel lower than the target dose for that cohort and a subsequent utomilumab infusion but experienced a DLT within 28 days after utomilumab infusion.
  No participants were enrolled in Phase 1: Cohort 5, so data is not available for them.
Measure: Number; unit: percentage of participants
Groups:
- Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg: Participants received cyclophosphamide 500 mg/m^2/day intravenously (IV) and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-cluster of differentiation (CD)19 chimeric antigen receptor (CAR) transduced autologous T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells was administered. Participants also received utomilumab 30 mg on Day 1, IV infusion, once every 4 weeks (Q4W) for 6 months or until progressive Disease, whichever came first.
- Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg: Participants received cyclophosphamide 500 mg/m^2/day intravenously (IV) and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-cluster of differentiation (CD)19 chimeric antigen receptor (CAR) transduced autologous T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells was administered. Participants also received utomilumab 100 mg on Day 1, IV infusion, once every 4 weeks (Q4W) for 6 months or until progressive Disease, whichever came first.
- Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg: Participants received cyclophosphamide 500 mg/m^2/day intravenously (IV) and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-cluster of differentiation (CD)19 chimeric antigen receptor (CAR) transduced autologous T cells/kg on Day 0. For participants weighing ≥ 100 kg, a maximum flat dose of axicabtagene ciloleucel at 2 x 10^8 anti-CD19 CAR T cells was administered. Participants also received utomilumab 200 mg on Day 1, IV infusion, once every 4 weeks (Q4W) for 6 months or until progressive Disease, whichever came first.
Arm/Group | Phase 1: Cohort 1: Axicabtagene Ciloleucel + Utomilumab 10 mg | Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg | Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg | Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3
percentage of participants | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 2: Complete Response (CR) Rate
Description: CR Rate: Percentage of participants with CR [complete metabolic response (CMR); complete radiological response (CRR)]. CMR: positron emission tomography (PET) 5-point scale (5-PS) scores of 1 (no uptake above background), 2 (uptake ≤ mediastinum), 3 (uptake > mediastinum but ≤ liver) with/without a residual mass); no new lesions; and no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow (BM). CRR: target nodes/nodal masses regressed to ≤ 1.5 cm in longest transverse diameter of lesion (LDi); no extralymphatic sites of disease; absent non-measured lesion (NMLs); organ enlargement regress to normal; no new sites; and bone marrow normal by morphology.
Time Frame: Up to 1 year
Population: Due to early termination of the study, Phase 2 of study was not conducted.
Groups:
- Phase 2: Axicabtagene Ciloleucel + Utomilumab: Participants were to receive cyclophosphamide and fludarabine conditioning chemotherapy followed by axicabtagene ciloleucel and utomilumab based on the dose/regimen selected to move forward from the Phase 1 portion of the study as recommended by the internal Safety Review Team.
  However, as the study was early terminated, no participants were enrolled in Phase 2 of this study.
Arm/Group | Phase 2: Axicabtagene Ciloleucel + Utomilumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Phase 1 and Phase 2: Objective Response Rate (ORR)
Description: ORR: Percentage of participants with CR [CMR;CRR] or PR [partial metabolic response (PMR); partial radiologic response (PRR)].CMR: PET 5PS scores of 1 (no uptake above background, 2 (uptake ≤ mediastinum), 3 (uptake>mediastinum but ≤ liver) with/without a residual mass; no new lesions; no evidence of FDG-avid disease in BM. CRR: target nodes/nodal masses regressed to ≤1.5 cm in LDi; no extralymphatic sites of disease; absent NMLs;organ enlargement regress to normal; no new sites; bone marrow morphology normal. PMR: scores 4 (uptake moderately > liver),5 (uptake markedly > liver, new lesions) with reduced uptake compared with baseline and residual mass; no new lesions; responding disease at interim/residual disease at end of treatment (EOT).PRR: ≥ 50% decrease in sum of the product of perpendicular diameters (SPD) of up to 6 target measurable nodes and extra-nodal sites;absent/normal, regressed, but no increase of NMLs; spleen regressed by > 50% in length beyond normal; no new sites.
Time Frame: From first infusion date of axicabtagene ciloleucel until first occurrence of CR or PR (maximum duration: 42.6 months)
Population: Participants in Safety Analysis Set were analyzed.
  No participants were enrolled in Phase 1: Cohort 5 and Phase 2, so data is not available for them.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: Cohort 1: Axicabtagene Ciloleucel + Utomilumab 10 mg | Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg | Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg | Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3
percentage of participants | 67 | 33 | 100 | 100

4. Secondary Outcome: Phase 1 and Phase 2: Duration of Response (DOR)
Description: DOR is time from first objective response (OR) to disease progression (PD)/death from any cause/up to last date known alive in the study. PD:score 4(uptake moderately>liver)/5(uptake markedly>liver and/or new lesions) with increase in intensity of uptake from baseline; new fluorodeoxyglucose (FDG)-avid foci consistent with lymphoma at interim/EOT assessment; new FDG-avid foci consistent with lymphoma rather than another etiology; new/recurrent FDG-avid foci in bone marrow; an individual node/lesion must be abnormal with: LDi >1.5 cm, increase by ≥50% from cross-product of LDi and perpendicular diameter (PPD) nadir, increase in LDi/shortest axis perpendicular to LDi from nadir, splenic length must increase by >50% of extent of its prior increase beyond baseline. If no prior splenomegaly, increase must be ≥2 cm from baseline; new/recurrent splenomegaly; new or clear progression of pre-existing NMLs; new lesion; new/recurrent bone marrow involvement. OR is defined in outcome measure 3.
Time Frame: From first documentation of CR or PR until first occurrence of PD or death from any cause or up to last date known alive in the study (maximum duration: 42.6 months)
Population: Participants in Safety Analysis Set were analyzed. DOR was assessed in participants with an objective response.
  No participants were enrolled in Phase 1: Cohort 5 and Phase 2, so data is not available for them.
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1: Cohort 1: Axicabtagene Ciloleucel + Utomilumab 10 mg | Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg | Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg | Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg
Number analyzed (Participants) | 2 | 1 | 3 | 3
months | 20.6 [18 to 23] | 22.1 [22.1 to 22.1] | 11.0 [5 to 24] | 17.3 [5 to 23]

5. Secondary Outcome: Phase 1 and Phase 2: Progression Free Survival (PFS)
Description: PFS is defined as the time from the axicabtagene ciloleucel infusion date to the date of PD per Lugano classification or death from any cause or up to last date known alive in the study. PD is defined in outcome measure 4.
Time Frame: From first infusion date of axicabtagene ciloleucel to the date of PD or death from any cause or up to last date known alive in the study (maximum duration: 43.5 months)
Population: as for outcome 3
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1: Cohort 1: Axicabtagene Ciloleucel + Utomilumab 10 mg | Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg | Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg | Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3
months | 23.8 [3 to 43] | 1.0 [1 to 35] | 12.0 [6 to 36] | 19.9 [6 to 24]

6. Secondary Outcome: Phase 1 and Phase 2: Overall Survival (OS)
Description: OS was defined as the time from axicabtagene ciloleucel infusion to the date of death from any cause or up to last date known alive in the study.
Time Frame: From first infusion date of axicabtagene ciloleucel to date of death from any cause or up to last date known alive in the study (maximum duration: 43.5 months)
Population: as for outcome 3
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1: Cohort 1: Axicabtagene Ciloleucel + Utomilumab 10 mg | Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg | Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg | Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3
months | 41.2 [5 to 43] | 35.1 [3 to 41] | 35.7 [30 to 36] | 24.4 [20 to 26]

7. Secondary Outcome: Phase 1 and Phase 2: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant in a clinical trial participant, which did not necessarily have a causal relationship with the treatment. TEAEs were defined as any worsening of a pre-existing medical condition that occurred on or after axicabtagene ciloleucel infusion or any AE with onset on or after axicabtagene ciloleucel infusion.
Time Frame: From first dose up to 30 days post last dose (maximum duration: 23.0 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: Cohort 1: Axicabtagene Ciloleucel + Utomilumab 10 mg | Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg | Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg | Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3
percentage of participants | 100 | 100 | 100 | 100

8. Secondary Outcome: Phase 1 and Phase 2: Percentage of Participants Experiencing Laboratory Toxicity Grade Shifts to Grade 3 or Higher Resulting From Increased Parameter Value
Description: Grading categories were determined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Grade 1: mild, Grade 2: moderate, Grade 3: severe or medically significant, Grade 4: life-threatening.
Time Frame: From first dose up to 30 days post last dose (maximum duration: 23.0 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: Cohort 1: Axicabtagene Ciloleucel + Utomilumab 10 mg | Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg | Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg | Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3
percentage of participants
  Glucose | 33 | 33 | 0 | 33
  Aspartate Aminotransferase | 0 | 0 | 0 | 33
  Bilirubin | 0 | 33 | 33 | 0
  Direct Bilirubin | 33 | 0 | 0 | 0
  Urate | 33 | 67 | 67 | 0
  Creatinine | 0 | 0 | 0 | 33
  Calcium | 0 | 67 | 0 | 0
  Magnesium | 0 | 0 | 33 | 33

9. Secondary Outcome: Phase 1 and Phase 2: Percentage of Participants Experiencing Laboratory Toxicity Grade Shifts to Grade 3 or Higher Resulting From Decreased Parameter Value
Description: as for outcome 8
Time Frame: From first dose up to 30 days post last dose (maximum duration: 23.0 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: Cohort 1: Axicabtagene Ciloleucel + Utomilumab 10 mg | Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg | Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg | Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3
percentage of participants
  Hemoglobin | 33 | 33 | 100 | 67
  Lymphocytes | 100 | 100 | 100 | 100
  Neutrophils | 100 | 100 | 100 | 100
  Platelets | 33 | 33 | 67 | 67
  Leukocytes | 100 | 100 | 100 | 100
  Calcium | 0 | 33 | 0 | 0
  Phosphate | 0 | 33 | 33 | 33
  Sodium | 33 | 0 | 0 | 33
  Potassium | 0 | 0 | 33 | 0

10. Secondary Outcome: Phase 1 and Phase 2: Pharmacokinetics: Peak Levels of Axicabtagene Ciloleucel in Blood
Description: Peak was defined as the maximum number of CAR T cells in blood measured after infusion.
Time Frame: Day 1 (Pre-utomilumab (UTO) Dose 1), Day 3 (Post-UTO Dose 1), Day 7, Day 10, Week 2, Week 3, Week 4 (Pre and Post-UTO Dose 2), Week 8 (Pre and Post-UTO Dose 3), Week 12 (Pre-UTO Dose 4), Week 16 (Pre-UTO Dose 5), Week 20 (Pre-UTO Dose 6), Week 24
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: cells/μL
Arm/Group | Phase 1: Cohort 1: Axicabtagene Ciloleucel + Utomilumab 10 mg | Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg | Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg | Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3
cells/μL | 11.99 [6.69 to 37.21] | 69.48 [36.98 to 996.87] | 149.40 [37.08 to 230.27] | 30.23 [16.63 to 103.38]

11. Secondary Outcome: Phase 1 and Phase 2: Pharmacodynamics: Peak Levels of Cytokines in Serum
Description: Peak is defined as the maximum post-baseline level of cytokine in the blood.
Time Frame: Baseline, Day 0, Day 7, Week 2, Week 4 (Pre and Post-UTO Dose 2)
Population: as for outcome 3
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 1: Cohort 1: Axicabtagene Ciloleucel + Utomilumab 10 mg | Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg | Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg | Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3
pg/mL
  CXCL10 | 763.60 [685.50 to 1794.80] | 2000.00 [1575.60 to 2000.00] | 865.60 [494.30 to 2000.00] | 2000.00 [616.90 to 2000.00]
  Granzyme B | 7.50 [6.60 to 19.20] | 42.20 [5.70 to 106.70] | 14.00 [4.30 to 44.90] | 13.60 [11.20 to 74.90]
  IFN-gamma | 40.30 [15.50 to 237.30] | 118.00 [76.20 to 303.30] | 216.60 [207.00 to 1876.00] | 761.90 [56.30 to 1876.00]
  IL-1 RA | 454.40 [339.90 to 1551.10] | 1100.00 [1006.00 to 1661.00] | 1578.00 [607.00 to 1639.00] | 2140.00 [901.00 to 9000.00]
  IL-2 | 0.90 [0.90 to 7.40] | 4.70 [3.50 to 8.60] | 27.70 [19.20 to 44.20] | 24.90 [5.50 to 87.10]
  IL-6 | 3.80 [1.60 to 26.40] | 111.20 [35.60 to 269.80] | 65.80 [19.50 to 897.40] | 976.00 [8.00 to 976.00]
  IL-8 | 31.70 [19.60 to 95.20] | 48.70 [23.20 to 63.30] | 121.60 [30.30 to 122.20] | 291.40 [36.80 to 750.00]
  TNF Alpha | 2.70 [1.70 to 6.00] | 7.30 [3.10 to 11.20] | 4.00 [3.50 to 8.70] | 4.10 [1.80 to 17.50]
  GM-CSF | 1.90 [1.90 to 1.90] | 1.90 [1.90 to 1.90] | 1.90 [1.90 to 5.90] | 7.50 [1.90 to 79.70]
  MCP-1 | 1063.30 [788.60 to 1143.10] | 1496.20 [415.00 to 1500.00] | 1500.00 [837.10 to 1500.00] | 1500.00 [956 to 1500.00]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Enrollment up to 43.5 months; Adverse events: From first dose up to 30 days post last dose (maximum duration: 23.0 months)
Description: All-cause mortality: Full Analysis Set defined as all enrolled participants who underwent leukapheresis.
  Adverse events: Safety Analysis Set defined as all participants treated with any dose of axicabtagene ciloleucel.
  No participants were enrolled in Phase 1: Cohort 5 and Phase 2, so data is not available for them.
Arm/Group | Phase 1: Cohort 1: Axicabtagene Ciloleucel + Utomilumab 10 mg | Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg | Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg | Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg
All-Cause Mortality (participants affected / at risk) | 3/5 | 2/4 | 1/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/3 | 1/3 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Cohort 1: Axicabtagene Ciloleucel + Utomilumab 10 mg (N=3) | Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg (N=3) | Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg (N=3) | Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Cohort 1: Axicabtagene Ciloleucel + Utomilumab 10 mg (N=3) | Phase 1: Cohort 2: Axicabtagene Ciloleucel + Utomilumab 30 mg (N=3) | Phase 1: Cohort 3: Axicabtagene Ciloleucel + Utomilumab 100 mg (N=3) | Phase 1: Cohort 4: Axicabtagene Ciloleucel + Utomilumab 200 mg (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0
Eyelid pain (Eye disorders) | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Catheter site pain (General disorders) | 1 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 2 | 0 | 3 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 3 | 3 | 2
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 1 | 1
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 2
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Viraemia (Infections and infestations) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 3 | 3
Platelet count decreased (Investigations) | 0 | 1 | 3 | 1
Respiratory syncytial virus test positive (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 2 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 1 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0
Headache (Nervous system disorders) | 3 | 3 | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 2 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 2 | 2 | 2 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT03704298/Prot_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/98/NCT03704298/SAP_001.pdf
  • Statistical Analysis Plan: Translational Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT03704298/SAP_002.pdf